CLINICAL TRIAL: NCT02641756
Title: In Depth Sampling and Subsequent Treatment Interruption to Identify the Anatomical Reservoir
Brief Title: HIV Sequencing After Treatment Interruption to Identify the Clinically Relevant Anatomical Reservoir
Acronym: HIV-STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIS 52777
Record Dates: First submitted 2015-12-09; First posted 2015-12-29 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2019-09

CONDITIONS: HIV
Keywords: HIV reservoir; phylogenetic analysis; sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Population (Experimental): This is a single arm study. The investigators will include 10 HIV positive patients under chronic CART (combined antiretroviral therapy).
  The intervention will consist on treatment interruption after in depth sampling under CART
  Interventions: Other: treatment interruption after in depth sampling under CART

INTERVENTIONS:
Other: treatment interruption after in depth sampling under CART — The participants will undergo in depth sampling under CART to characterise the HIV reservoir in different anatomical compartments. Subsequently an experimental viral rebound, by a brief therapy stop, will help us identify the clinically relevant viral reservoir by doing phylogenetic analysis on the rebounding virus and on the virus found in the different compartments under CART.

SUMMARY:
The main goal of this study is to identify and characterise the anatomical component of the replication competent HIV-1 (Human Immunodeficiency Virus-1) reservoir.

The investigators hypothesize that the clinically relevant HIV-1 reservoir is hiding in various but specific anatomic compartments and is able to rebound when therapy is stopped.

This reservoir is probably smaller than the HIV-1 reservoir hiding in the blood but could be more transcriptional active because of its specific environment, possibly influenced by lower concentrations of the antiretroviral therapy.

The current proposal will, for the first time, identify the source of the viral reservoir by phylogenetically backtracking the viral genome of the rebounding virus to the sequences of viral DNA (DeoxyriboNucleic Acid) in different anatomical compartments. The subsequent characterization of the viral reservoir markers (size, integration sites, methylation profile, stimulation and inhibition assays) will enable us to understand how this viral rebound occurred.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection, subtype B
* Able and willing to provide written informed consent
* Age = or >18 years < 65 years
* Nadir CD4 (cluster of differentiation 4) count >=300/µl. Cluster of differentiation 4 (CD4) count at screening > 500/μl
* Patient should take antiretroviral therapy (ART) for at least 2 years with no changes in the ART for at least 90 days prior to study entry. Patients should be on an integrase inhibitor + 2 nucleoside analogs based regimen or PI based regimen.
* Patient should have a viral load < 20 copies/ml determined by CobasTaqMan HIV-1 test v2.0 assay for at least 2 years. (Occasional "blips" will be permitted) (A blip is defined as an intermittent viremic episode with a viral load above detection level but below 200 copies/ml and a return to an undetectable level in a next control, if more than six months prior to the study entry)
* Last viral load undetectable
* Ability to attend the complete schedule of assessments and patient visits. Ability and willingness to have blood and tissue samples collected and stored indefinitely and used for various research purposes. Women of childbearing potential or their partner should use double barrier contraception during the study. Females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy, or bilateral oophorectomy and/or bilateral salpingectomy), will need a negative serum or urine pregnancy test within 48 hours prior to study entry.

Note: Acceptable documentation of hysterectomy and bilateral oophorectomy, bilateral salpingectomy, tubal micro-inserts, partner who has undergone vasectomy, and menopause is participant-reported history. All participants must agree not to participate in the conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, or in vitro fertilization). Participants must agree to use barrier protection for all sexual activity and if participating in sexual activity that could lead to pregnancy, the participant/partner must use at least two reliable forms of contraceptives (condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an intra-uterine device (IUD); or hormone-based contraception) during the study.

Exclusion Criteria:

* Previous or current history of opportunistic infection. (AIDS defining events as defined in category C of the Center for Disease Control and Prevention (CDC) clinical classification).
* History of resistance to antiretroviral drugs, documented by genotyping.
* Hepatitis B surface antigen positive or Hepatitis B virus (HBV) viral load positive in the past and no evidence of subsequent seroconversion (=HBV antigen or viral load negative and positive HBV surface antibody).
* Hepatitis C virus (HCV) antibody positive result within 60 days prior to study entry or, if the HCV antibody result is negative, a positive HCV RNA (Ribonucleic Acid) result within 60 days prior to study entry
* Significant risk of HIV superinfection during treatment interruption.
* Current or known history of cardiomyopathy or significant ischemic or cerebrovascular disease.
* History of HIV-related thrombocytopenia.
* Active renal disease (defined as a glomerular filtration rate (calculated by Cockcroft Gault equation) below 50ml/min or the presence of HIV-associated nephropathy (HIVAN) in the past medical history.
* Current or known history of cancer (with the exception of in situ cervix carcinoma or squamous cell carcinoma of the skin) within five years prior to screening.
* Pregnancy or breastfeeding.
* Any conditions, including psychiatric and psychological disorders, which will in the opinion of the investigator interfere with the trial conduct or safety of the participant.
* Previous participation in a trial evaluating an immune modulating agent
* Abnormal laboratory tests results at screening:

  1. Confirmed Hemoglobin <11g/dl for women and <12 g:dl for men
  2. Confirmed platelet count < 100000/l
  3. Confirmed neutrophil count <1000/μl
  4. Confirmed aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2x Upper Limit of Normal (ULN)

The following treatment will be prohibited three months before screening and during the course of the study:

1. immunosuppressive drugs (inclusive corticosteroids) with the exception of drugs used for topical use.
2. Immunomodulatory drugs including but not limited to Granulocyte colony stimulating factors, Granulocyte-monocyte stimulating factor, interleukin 2, 7 & 15.

   * Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
   * Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 60 days prior to entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Phylogenetic analysis of the virus found in the different compartments under treatment and of the virus in the plasma at viral rebound. | 24 months
  Genetically link the viral reservoir in different anatomical reservoirs to the rebounding virus found in the plasma after therapy-stop by doing phylogenetic analysis. This will be done by a method called single proviral sequencing.

SECONDARY OUTCOMES:
Number of patients with adverse events that are related to the study intervention, graded according to NCI CTCAE Version 4.0 | 24 months
  Assess safety of the experimental treatment interruption for future clinical trials. Confirmation of the safety of a treatment interruption strategy in selected patients will be based on the number and intensity of AEs (adverse events) graded according to the NCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE) on a five-point scale (Grade 1 to 5: Mild, Moderate, Severe, Life-threatening and Death).
The severity of adverse events that are related to the study intervention, graded according to NCI CTCAE Version 4.0 | 24 months
  Assess safety of the experimental treatment interruption for future clinical trials. Confirmation of the safety of a treatment interruption strategy in selected patients will be based on the number and intensity of AEs (adverse events) graded according to the NCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE) on a five-point scale (Grade 1 to 5: Mild, Moderate, Severe, Life-threatening and Death).
Psychological effects of treatment interruption | 24 months
  The investigators will evaluate psychological effects of the treatment interruption by a questionnaire.
Evaluation of the reservoir replenishment by quantifying the viral reservoir under combined antiretroviral therapy (CART) in various anatomic compartments.(Total HIV DNA, integrated HIV DNA, Cell-associated-HIV RNA). | 24 months
  Assessment of the viral reservoir magnitude prior and after treatment interruption by quantification of viral reservoir by ultrasensitive polymerase chain reaction (PCR) methods.
Evaluation of the reservoir replenishment by quantifying the viral reservoir under combined antiretroviral therapy (CART) in various anatomic compartments.(viral outgrowth assay). | 24 months
  Assessment of the viral reservoir magnitude prior and after treatment interruption by replication competence of the virus by reactivation assays.
Therapeutic drug monitoring assessed by drug concentrations measured in the different compartments | 24 months
  assess drug concentrations in different compartments and its significance in maintaining the HIV reservoir
Assessment of the kinetics of HIV viral load rebound after treatment interruption based on the repetitive plasma viral load measurements. | 6 months
  The kinetics will be on the plasma viral load (expressed in copies/ml) measured two-weekly until viral rebound.

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, Prof, Principal Investigator — UZ Gent - U Gent
Locations (1):
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cole B, Lambrechts L, Boyer Z, Noppe Y, De Scheerder MA, Eden JS, Vrancken B, Schlub TE, McLaughlin S, Frenkel LM, Palmer S, Vandekerckhove L. Extensive characterization of HIV-1 reservoirs reveals links to plasma viremia before and during analytical treatment interruption. Cell Rep. 2022 Apr 26;39(4):110739. doi: 10.1016/j.celrep.2022.110739. PMID 35476994
- [Derived] De Scheerder MA, Van Hecke C, Zetterberg H, Fuchs D, De Langhe N, Rutsaert S, Vrancken B, Trypsteen W, Noppe Y, Van Der Gucht B, Pelgrom J, Van Wanzeele F, Palmer S, Lemey P, Gisslen M, Vandekerckhove L. Evaluating predictive markers for viral rebound and safety assessment in blood and lumbar fluid during HIV-1 treatment interruption. J Antimicrob Chemother. 2020 May 1;75(5):1311-1320. doi: 10.1093/jac/dkaa003. PMID 32053203
- See also: publication — https://doi.org/10.1016/j.chom.2019.08.003

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT02641756/Prot_SAP_000.pdf